CLINICAL TRIAL: NCT00923390
Title: Phase 1/2 Study of Metastatic Renal Cancer Using T-Cells Transduced With a T-Cell Receptor Which Recognizes TRAIL Bound to the DR4 Receptor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090092; 09-C-0092; NCT00870389 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2012-08-24

CONDITIONS: Renal Cancer; Kidney Cancer
Keywords: Renal Cancer; Immunotherapy; Clinical Response; Toxicity; Gene Therapy; Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — aldesleukin; Cyclophosphamide; fludarabine

INTERVENTIONS:
Genetic: 2G-1 TCR Retroviral Vector-Transduced lyn
Drug: Aldesleukin
Drug: Cyclophosphamide
Drug: Fludarabine
Drug: (PG13-A(F/K-F-SGSG-T2a-B (opt) (2G-1 TCR) retroviral vector-transduced lymphocyte

SUMMARY:
Background:

* An experimental cancer treatment procedure involves taking a patient s own tumor or blood cells, modifying them with a gene that targets proteins on the surface of tumor cells, and growing those cells in a laboratory. The modified cells are then given back to the patient by intravenous (IV) transfusion, in the hope that the new cells will attack and destroy the cancer cells without harming healthy tissue.
* This procedure has been used for melanoma patients, and researchers are now attempting to use this treatment for patients with renal (kidney) cancer. In the laboratory, this attack kills nearly all kidney cancers tested, but not normal tissues. However, the effectiveness and possible side effects of this treatment are still being studied.

Objectives:

* To find out if cells modified to target DR4 and TRAIL (two proteins found on the surface of many kidney tumors) are effective in treating kidney cancer.
* To determine the maximum tolerated dose (the highest dose that does not cause unacceptable side effects) of the modified cells.

Eligibility:

* Patients 18 years of age and older with metastatic renal cancer whose disease has not responded to standard treatment.
* Patients will be divided into two study branches: Arm A for those who will be receiving modified cells from their biopsied tumor, and Arm B for those who will be receiving their own modified white blood cells.

Design:

* Five-stage treatment process, outpatient for stages 1 and 5 and inpatient for stages 2 through 4:
* Work-up (1 to 2 weeks): Physical examination, heart and lung function tests, imaging tests, blood and/or tumor samples taken.
* IV chemotherapy (1 week): Cyclophosphamide and fludarabine to prepare for the new cell infusion.
* IV cell infusion and treatment with IL-2 to support the modified cells (4 days).
* Recovery (1 to 2 weeks): Recover from effects of chemotherapy and infusion.
* Follow-up (every 1 to 6 months): Return to clinic for physical exam, review of side effects, other tests.
* Follow-up evaluations will continue to determine the success of the treatment.
* Evaluations during the treatment period:
* Physical examination, including vital signs and body weight checks, and pregnancy test for women who can become pregnant.
* Blood and urine tests.
* Disease evaluation and monitoring on both inpatient and outpatient basis.
* Because researchers do not know the long-term side effects of gene therapy, patients will be asked to participate in long-term follow up for up to 15 years. The follow-up will involve yearly physical exams and medical history, and blood collection (3, 6 and 12 months after treatment, and every year after that).

DETAILED DESCRIPTION:
Background:

* The clinical administration of tumor-reactive T-cells grown in vitro is a highly active therapy for patients with metastatic melanoma in experimental protocols when they are combined with preparative lymphodepleting chemotherapy and systemic IL-2.
* We cloned a novel T-cell from the blood of a patient with renal cell cancer (RCC), which recognizes nearly all human renal cancer lines irrespective of MHC haplotype.
* The alpha sign and beta sign chain of T-cell receptor from this clone, 2G-1, can be introduced into human lymphocytes by retroviral transduction and confers this same recognition of RCC.
* This TCR was found to recognize TNF-related apoptosis inducing ligand (TRAIL) bound to its receptor DR4.
* Both TRAIL and agonist antibodies to DR4 have tumor specificity and are in current clinical trials for cancer.
* Two amino acid modifications of the native TCR greatly augmented its recognition of RCCs without altering background reactivity.

Objectives:

* Primary:

  * Determine if the administration of T-cells retrovirally transduced with the 2G-1 TCR, with preparative chemotherapy and IL-2, can cause the regression of metastatic RCC.
  * To identify the maximum tolerated dose (MTD) for cells incorporating a TCR in PBL and in TIL.
* Secondary:

  * Determine the toxicities of these T-cells administered in the above fashion.
  * Determine TCR and vector presence in the post treatment phase.

Eligibility:

* Patients with measurable metastatic clear cell renal cancer who have previously received at least one systemic standard care regimen and have progressed or be found to be intolerant of standard therapies.
* Patients must be eligible for high-dose IL-2.
* Patients must not have active or clinically symptomatic CNS metastases within the previous 3 months.
* Patients must have acceptable hematopoietic and major organ function as determined by laboratory and/or functional testing.

Design:

* A phase I-II dose escalating protocol with 2 arms. Patients in Arm A will receive peripheral blood lymphocytes transduced with the 2G-1 TCR; patients in Arm B will receive renal TIL transduced with the 2G-1 TCR. Arm B will begin after a safe dose has been defined in Arm A.
* Once MTD has been established for each arm, up to 24 patients will be enrolled in each arm of the phase II stage.
* Patients will receive a nonmyeloablative but lymphocyte-depleting preparative regimen consisting of cyclophosphamide and fludarabine followed in one to four days by IV infusion of their transduced cells and subsequent IV aldesleukin administration.
* Up to 106 patients may be enrolled over 3-4 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Measurable metastatic clear cell renal cancer. Histologic diagnosis will be confirmed by the Laboratory of Pathology at the NCI.
  2. Patients must have previously received at least one systemic standard care regimens and have progressed or be found to be intolerant of standard therapies.
  3. Greater than or equal to 18 years of age.
  4. Willing to sign a durable power of attorney
  5. Able to understand and sign the Informed Consent Document
  6. Clinical performance status of ECOG 0 or 1.
  7. Life expectancy of greater than three months.
  8. Patients of both genders must be willing to practice birth control during and for four months after receiving the preparative regimen.
  9. Serology:

     1. Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immunecompetence, and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
     2. Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.
     3. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
  10. Hematology:

      1. Absolute neutrophil count greater than or equal to 1000/mm3 without the support of filgrastim.
      2. WBC greater than or equal to 3000/mm3.
      3. Platelet count greater than or equal to 100,000/mm3.
      4. Hemoglobin greater than or equal to 8.0 g/dl.
  11. Chemistry:

      1. Serum ALT/AST less or equal to 2.5 times the upper limit of normal.
      2. Serum creatinine less than or equal to 1.6 mg/dl.
      3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert s Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  12. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for alopecia or skin rash, which must have recovered to a grade 2 or less).
  13. Patients who have previously received anti-CTLA4 antibody must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
2. Active systemic infections; coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system; myocardial infarction; cardiac arrhythmias; obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
5. Concurrent systemic steroid therapy
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. History of coronary revascularization or ischemic symptoms
8. Documented LVEF less than or equal to 45%. LVEF will be evaluated in patients with:

   1. History of ischemic heart disease, chest pain, or clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
   2. Age greater than or equal to 60 years old
9. Documented FEV1 less than or equal to 60% predicted. Screening pulmonary function testing will be done in patients with:

   1. A prolonged history of cigarette smoking (20 pk/year of smoking, who have not quit within the past 2 years).
   2. Symptoms of respiratory dysfunction
10. Patients who have a history of more than two CNS metastases.
11. Patients who have any CNS lesion that is symptomatic, greater than 1 cm in diameter or shows significant surrounding edema on MRI scan will not be eligible until they have been treated and demonstrated no clinical or radiologic CNS progression for at least 2 months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-03-02; Primary Completion 2012-08-24 (Actual); Study Completion 2012-08-24 (Actual)

PRIMARY OUTCOMES:
Determine if the administration of T-cells retrovirally transduced with the 2G-1 TCR, with preparative chemotherapy and IL-2, can cause the regression of metastatic RCC, and to identify the maximum tolerated dose for the 2G-1 TCr transduced cell...

SECONDARY OUTCOMES:
Determine the toxicities of these T-cells administered in the above fashion, and to determine TCR and vector presence in the post treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: James C Yang, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Motzer RJ, Michaelson MD, Rosenberg J, Bukowski RM, Curti BD, George DJ, Hudes GR, Redman BG, Margolin KA, Wilding G. Sunitinib efficacy against advanced renal cell carcinoma. J Urol. 2007 Nov;178(5):1883-7. doi: 10.1016/j.juro.2007.07.030. Epub 2007 Sep 17. PMID 17868732
- [Background] Bukowski RM, Kabbinavar FF, Figlin RA, Flaherty K, Srinivas S, Vaishampayan U, Drabkin HA, Dutcher J, Ryba S, Xia Q, Scappaticci FA, McDermott D. Randomized phase II study of erlotinib combined with bevacizumab compared with bevacizumab alone in metastatic renal cell cancer. J Clin Oncol. 2007 Oct 10;25(29):4536-41. doi: 10.1200/JCO.2007.11.5154. Epub 2007 Sep 17. PMID 17876014
- [Background] Klapper JA, Downey SG, Smith FO, Yang JC, Hughes MS, Kammula US, Sherry RM, Royal RE, Steinberg SM, Rosenberg S. High-dose interleukin-2 for the treatment of metastatic renal cell carcinoma : a retrospective analysis of response and survival in patients treated in the surgery branch at the National Cancer Institute between 1986 and 2006. Cancer. 2008 Jul 15;113(2):293-301. doi: 10.1002/cncr.23552. PMID 18457330